CLINICAL TRIAL: NCT05823675
Title: A Phase 1 Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Clinical Activity of Itolizumab in Subjects With Newly Diagnosed Acute Graft Versus Host Disease
Brief Title: Safety and Clinical Activity of Itolizumab in aGVHD
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Biotech Pharmaceutical Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BPL-ITO-aGVHD-1
Record Dates: First submitted 2023-03-16; First posted 2023-04-21 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-04

CONDITIONS: Acute Graft Versus Host Disease
MeSH Terms: interventions — itolizumab; Methylprednisolone; Methylprednisolone Hemisuccinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Itolizumab Dose Level 1 (Experimental): Itolizumab of 25 mg administered by intravenous infusion every 2 weeks for a total of 5 doses.
  Interventions: Drug: Itolizumab; Drug: Methylprednisolone
- Itolizumab Dose Level 2 (Experimental): Itolizumab of 50 mg administered by intravenous infusion every 2 weeks for a total of 5 doses.
  Interventions: Drug: Itolizumab; Drug: Methylprednisolone
- Itolizumab Dose Level 3 (Experimental): Itolizumab of 100 mg administered by intravenous infusion every 2 weeks for a total of 5 doses.
  Interventions: Drug: Itolizumab; Drug: Methylprednisolone
- Itolizumab Dose Level 4 (Experimental): Itolizumab of 150 mg administered by intravenous infusion every 2 weeks for a total of 5 doses.
  Interventions: Drug: Itolizumab; Drug: Methylprednisolone

INTERVENTIONS:
Drug: Itolizumab — Subjects will receive Itolizumab concomitant within 72 hours of systematic Corticosteroids.
  Other Names: T1h
Drug: Methylprednisolone — Methylprednisolone will be taperred as required
  Other Names: Methylprednisolone Sodium Succinate

SUMMARY:
To evaluate the safety, tolerability, PK, PD, and clinical activity of Itolizumab in subjects with Newly diagnosed Acute Graft Versus Host Disease(aGVHD).

DETAILED DESCRIPTION:
The study will enroll approximately 44 subjects in three parts:

Part 1 is an open label 3+3 single dose escalation phase and will enroll approximately 30 subjects with aGVHD across 4 cohorts, where subjects will receive Itolizumab administered intravenously for 1 dose.

Part 2 is an open label phase and subjects from part 1 will receive Itolizumab administered intravenously every two weeks for a total of 4 doses.

Part 3 is a randomized phase and will enroll approximately 14 additional subjects, randomized in a 1:1 ratio to one of the 2 recommended doses provided by Part 1 and Part 2. Subjects will receive Itolizumab administered intravenously every two weeks for a total of 5 doses.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject at least 18 years of age.
* Has received allogeneic hematopoietic stem cell transplantation (allo-HSCT).
* Clinical diagnosis of Grade II-IV aGVHD per MAGIC guideline requiring systemic immune suppressive therapy.
* Initiation of systemic steroids therapy ≤ 72 hours.
* Negative result of serum HCG within 72 hours before enrollment for female with potential fertility.
* Have a life expectancy of 10 weeks or more.
* Able to understand and comply with the planned procedure as required by the protocol, and sign a written informed consent form (ICF).

Exclusion Criteria:

* Has received more than 1 allo-HSCT.
* Presence of morphologic relapsed primary malignancy, treatment for relapse after alloHSCT was performed, or requirement for rapid immunosuppressive treatment withdrawal for early malignancy relapse.
* Evidence of graft failure based on cytopenia(s), and as determined by the investigator.
* Evidence of post-transplant lymphoproliferative disease.
* Any prior therapy for acute GVHD, except for alloHSCT prophylaxis regimens or systemically administered corticosteroids.
* aGVHD induced by donor lymphocyte infusion(DLI).
* Clinically or suspected diagnosed of cGVHD or overlap syndrome.
* Unresolved toxicity or complications due to allo-HSCT,other than aGVHD.
* Any clinical or laboratory abnormalities that is likely to negatively affect the reliability of the study safety data, as determined by the investigator.
* Presence of any uncontrolled active infections, which was defined as hemodynamic instability due to sepsis or worsening of new symptoms, signs, or imaging findings due to infection.
* Presence of any uncontrolled and active infections.
* Presence of active and uncontrolled viral infections at screening.
* History of active tuberculosis within 6 months prior to screening or negative result of interferon-gamma release assay at screening.
* History of class III or IV congestive heart failure per New York Heart Association, clinically significant or uncontrolled unstable angina or myocardial infarction, cerebrovascular accident, or pulmonary embolism within 6 months prior to screening.
* Severe impaired renal function at screening (serum creatinine > 1.5 ULN or creatinine clearance < 30mL/min).
* Presence of persistent bilirubin abnormalities induced by hepatic sinusoidal obstruction, hepatic veno-occlusive disease, non-GVHD or progressive organ dysfunction at screening.
* Serum ALT and AST > 4 ULN at screening.
* Absolute lymphocyte count < 0.5×109/L at screening.
* Any major surgical procedures performed within 4 weeks prior to screening, that is likely to negatively affect the evaluation of the study safety data, as determined by the investigator.
* Any malignant tumor other than the transplanted tumor within 5 years before screening.
* Suspected allergic to the experimental drug product or any of its excipients.
* Currently pregnant, breastfeeding,or planning to become pregnant or not using reliable method to avoid pregnancy during study and within 3 months after the last study treatment.
* As determined by the investigator, any medical, psychiatric, or other condition or circumstance that is likely to negatively affect the reliability of the study data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2023-05-19 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment Emergent Adverse Events | Study Day 85
  Number of subjects with treatment-related adverse events as assessed by the Common Terminology Criteria for Adverse Events (CTCAE) V5.0

SECONDARY OUTCOMES:
Time to maximum Itolizumab serum concentration, Tmax | Study Day 85
  Time to maximum Itolizumab serum concentration
Maximum Itolizumab serum drug concentration, Cmax | Study Day 85
  Maximum Itolizumab serum drug concentration
Minimum Itolizumab serum drug concentration, Cmin | Study Day 85
  Minimum Itolizumab serum drug concentration
Total Itolizumab exposure across time, AUC | Study Day 85
  Total Itolizumab exposure across time, AUC
Half life of Itolizumab, t1/2 | Study Day 85
  Half life of Itolizumab
Volume of distribution of Itolizumab, Vd | Study Day 85
  Volume of distribution of Itolizumab
Clearance, Cl | Study Day 85
  Clearance
CD6 receptor expression levels on T cells | Study Day 85
  CD6 receptor expression levels
T cell subsets | Study Day 85
  T cell subsets
Inflammatory Markers | Study Day 85
  Including but not limited to:IL-2, IL-6, IL-8, IL-17, IFN-γ, TNF-α, CRP, TNFR1, ST2, REG3α, Elafin
Overall Response Rate (ORR) | Study Day 337
  Percentage of subjects demonstrating a CR or PR.
Nonrelapse Mortality(NRM) Rate | Study Day 337
  Proportion of subjects who died due to causes other than malignancy relapse
cGVHD rate | Study Day 337
  Percentage of subjects demonstrating of cGVHD
Dose Reduction in Systemic Steroid Use | Study Day 337
  Change from Baselinein Dose of Systemic Steroid Use
Incidence of ADA | Study Day 85
  Precentage of subjects presenting anti-drug antibody

CONTACTS AND LOCATIONS:
Overall Officials: Erlie Jiang, Principal Investigator — Chinese Academy of Medical Sciences
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Chinese Academy of Medical Sciences & Peking Union Medical College, Tianjin, China

IPD SHARING:
Plan to Share IPD: No